CLINICAL TRIAL: NCT01379755
Title: Study of Compare Mid-flexion Stability and Clinical Outcomes in Single-radius Femoral Design or Multi-radius Femoral Design.
Brief Title: Comparison of Stability and Outcomes in Single-radius Femoral Component for Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: JK Seon, Center for Joint Disease, Chonnam National University Hwasun Hospital
Other Study IDs: singleradius; singleradius2 (Other: Chonnam National University Hwasun Hospital)
Record Dates: First submitted 2011-06-08; First posted 2011-06-23 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis
Keywords: stability; single-radius; multi-radius; total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a comparison of the functional results and Varus-Valgus Stability in Single-radius versus Multi-radius Femoral Component for Total Knee Arthroplasty.

DETAILED DESCRIPTION:
Recently, femoral designs based on a sagittal single radius were designed to allow better mid-flexion stability and extensor function after total knee arthroplasty. The purpose of this study was to compare mid-flexion stability and clinical outcomes in patients that received TKA using either a single-radius femoral design or multi-radius femoral design.

ELIGIBILITY:
Inclusion Criteria:

* followed for a minimum of two years.

Exclusion Criteria:

* Not followed for a minimum of two years.

Ages: 48 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 56 total knee arthroplasties(TKAs) with a single-radius femoral design (Scorpio NRG) (single-radius(SR) group) and 59 total knee arthroplasties(TKAs) with multiradius femoral design (NexGen CR) (multi-radius(MR) group)
Sampling Method: Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Keun Seon, Professor, Study Director — Center for Joint Disease, Chonnam National University Hwasun Hospital, Jeonnam, Korea
Locations (1):
- Center for Joint Disease, Chonnam National University Hwasun Hospital, Hwasun-Gun, Jeollanam-do, South Korea